CLINICAL TRIAL: NCT05501977
Title: Retrospective Analysis of Factors Affecting Chronic Postoperative Pain After Thoracotomy
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Associate Professor, Ankara University
Other Study IDs: 10483751
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Chronic Pain Syndrome; Thoracotomy
MeSH Terms: interventions — Thoracotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with chronic pain after thoracotomy: patients with chronic pain after thoracotomy
  Interventions: Procedure: thoracotomy
- patients without chronic pain after thoracotomy: patients without chronic pain after thoracotomy
  Interventions: Procedure: thoracotomy

INTERVENTIONS:
Procedure: thoracotomy — thoracic surgery for pulmonary diseases

SUMMARY:
The aim of this retrospective study is to determine the factors affecting the development of chronic pain in patients with thoracotomy in the Thoracic Surgery Operating Rooms of İbn-i Sina Hospital. By identifying these factors, it is aimed to apply the necessary treatments to prevent the development of chronic pain and to improve patient outcomes.

DETAILED DESCRIPTION:
The study included 229 patients ASA 1, 2 and 3, 18 years of age and older, who underwent elective thoracotomy in Ankara University İbn-i Sina Hospital, Thoracic Surgery operating room between 01.01.2016 and 31.12.2020. The medical files and electronic records of the patients were scanned from the system. Age, gender, weight, ASA score, smoking, comorbidities (hypertension, diabetes), drug use, malignancy, chemotherapy history, radiotherapy history, intraoperative and postoperative analgesia method, duration of acute pain, type of surgery, duration of surgery, duration of anesthesia, rib resection, number of chest tubes and duration time, time to apply to the pain clinic, and the analgesic method applied were recorded.

ELIGIBILITY:
Inclusion Criteria:

* asa 1,2 and 3
* 18 year of age and older
* underwent elective thoracotomy

Exclusion Criteria:

* ASA 4 and 5, emergency or trauma thoracotomy, patients with malignancy infiltrating the chest wall, more than one thoracotomy performed, patients whose cardiovascular or cerebrovascular or musculoskeletal system was affected at a level that would affect their daily activities after surgery, and patients with insufficient data for various reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent elective thoracotomy ASA 1, 2 and 3, 18 years of age and older in Ankara University İbn-i Sina Hospital, Thoracic Surgery operating room between 01.01.2016 and 31.12.2020 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
number of patients who had chronic pain after thoracotomy | 3 months
  number of patients who had chronic pain after thoracotomy

SECONDARY OUTCOMES:
type of analgesic | 3 months
  analgesic methods used for acute postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, Study Director — Ankara University
Locations (1):
- Cigdem Yildirim Guclu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided